CLINICAL TRIAL: NCT04994015
Title: Parkinson's Foundation PD GENEration Genetic Registry
Status: Recruiting | Type: Observational
Sponsor: Parkinson's Foundation (Other)
Collaborators: Indiana University (Other); Fulgent Genetics (Unknown); The Parkinson Study Group (Network)
Responsible Party: Sponsor
Other Study IDs: PDGENE-PF
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Parkinson's Disease
Keywords: Genetics; Genetic Counseling; Whole Genome Sequencing
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples With DNA — Isolated DNA from buccal swab or whole blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Lab Assay for seven genetic variants for Parkinson's Disease — Counseling provided to participant by site clinician/physician/genetic counselor.

SUMMARY:
Development of a central repository for PD-related genomic data for future research.

DETAILED DESCRIPTION:
The purpose of this study is to develop a central repository for PD-related genomic data by individuals who consent to deposit their data and bank their residual DNA obtained through clinical genetic testing for future research use.

ELIGIBILITY:
Inclusion Criteria:

* Study Population 1: PWP (open for recruitment)

  1. Meet Movement Disorder Society (MDS) Clinical Diagnostic Criteria for Parkinson's Disease: probable diagnosis.
  2. Willingness to undergo genetic testing, and choose to be informed of genetic testing results for GBA, LRRK2 and 5 additional PD related genes (SNCA, VPS35, PRKN, PINK-1, PARK7).
  3. Capacity to give full informed consent in writing or electronically, and have read and signed the informed consent forms (ICFs) based on site clinician's determination.
  4. Able to perform study activities (including completion of either online, in-person or paper surveys).

Study Population 2: People at risk of developing PD (not open for recruitment)

1. Family members of Study Population 1 may be invited to participate in the study if confirmatory genetic testing is deemed necessary by the genetic testing laboratory.

Exclusion Criteria:

1. Diagnosis of an atypical parkinsonian disorder (i.e., multiple system atrophy, progressive supranuclear palsy, dementia with Lewy bodies, corticobasal syndrome), including that due to medications, metabolic disorders, encephalitis, cerebrovascular disease, or normal pressure hydrocephalus.
2. Individuals who have received a blood transfusion within the past 3 months.
3. Individuals who have active hematologic malignancies such as lymphoma or leukemia.
4. Individuals who have had a bone marrow transplant within the past 5 years.
5. Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any person with probable diagnosis of Parkinson's disease according to the Movement Disorders Society criteria.
Sampling Method: Non-Probability Sample
Enrollment: 25000 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Parkinson's related genetic mutations in an convenience cohort | 6 months
  Identify people with Parkinson's who have genetic mutations to advance basic science and clinical research.
Educating people with Parkinson's of their genetic mutation status through genetic testing and counseling | 6 months
  People who are informed of their genetic status may be empowered to learn more about their disease and participant in clinical research.

CONTACTS AND LOCATIONS:
Overall Officials: James Beck, PhD, Principal Investigator — Parkinson's Foundation; Roy N Alcalay, MS, MD, Principal Investigator — Tel Aviv Sourasky Medical Center, Columbia University Irving Medical Center
Locations (56):
- United States (54):
  - University of Alabama Birmingham, Birmingham, Alabama
  - MD First Research, Chandler, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of Arkansas, Fayetteville, Arkansas
  - University of California San Diego (UCSD), La Jolla, California
  - University of California Los Angeles, Los Angeles, California
  - University of California San Francisco (UCSF), San Francisco, California
  - University of Colorado Anschutz, Aurora, Colorado
  - Hartford Healthcare, Hartford, Connecticut
  - Aventura Neurology - Visionary Investigators Network, Aventura, Florida
  - Parkinson's Disease & Movement Disorder Center of Boca Raton, Boca Raton, Florida
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Cleveland Clinic Weston, Weston, Florida
  - Morehouse College, Atlanta, Georgia
  - The Queen's Health System, Honolulu, Hawaii
  - University of Illinois-Chicago, Chicago, Illinois
  - Rush University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas, Lawrence, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Louisiana State University, Shreveport, Louisiana
  - Johns Hopkins, Baltimore, Maryland
  - University of Maryland, College Park, Maryland
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - BMC Community Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Struthers Parkinson's Center - HealthPartners Park Nicollet, Golden Valley, Minnesota
  - Rutgers University, New Brunswick, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - New York University, New York, New York
  - Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Atrium Health, Charlotte, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Texas at San Antonio, San Antonio, Texas
  - Intermountain Health, Murray, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Evergreen Health, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Toronto Western Hospital, Toronto, Ontario, Canada
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

DOCUMENTS (1):
  • Informed Consent Form (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/15/NCT04994015/ICF_000.pdf